CLINICAL TRIAL: NCT04274140
Title: Maternal Obesity and Offspring Neurodevelopment: the MOON Study
Brief Title: Maternal Obesity and Offspring Neurodevelopment
Acronym: Moon
Status: Active, not recruiting | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 239304
Record Dates: First submitted 2019-11-13; First posted 2020-02-18 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obese Pregnant Women: obese, BMI 30-50
- Normal weight pregnant women: normal weight, BMI 18.5-25

SUMMARY:
Our goals are to characterize the effects of maternal obesity during pregnancy on infant brain development, reveal the neurodevelopmental consequences, and identify possible mechanisms causing these effects. Our overall hypothesis is that maternal obesity during pregnancy exposes the fetus to an inflammatory environment that affects infant brain structural and functional development and consequently neurodevelopmental outcomes. To test this hypothesis, the investigators will recruit normal-weight and obese pregnant women, examine inflammatory markers associated with obese pregnancy, and correlate them with offspring's brain development evaluated using quantitative MRI methods and outcomes evaluated using neurodevelopmental tests.

DETAILED DESCRIPTION:
About one third of all women of reproductive age in the US are obese (body mass index [BMI] ≥ 30). Recent studies show that children born to mothers who were obese while pregnant may have lower cognitive performance and higher risk of developing neurodevelopmental conditions. The goal of this study is to see 1) if there are negative effects of maternal obesity during pregnancy on newborn's brain development; 2) if these effects on brain development persist to age 1 & 2 years, and if there are changes in neurodevelopmental outcomes associated with maternal obesity; and 3) if inflammation in pregnant women associated with maternal obesity is one of the main reasons for the brain changes in offspring. The investigators will recruit pregnant women from early pregnancy who are either obese or normal weight and are otherwise healthy. The Investigators will measure their weight, body fat percentage, blood inflammation markers, family environment, what the participants normally eat, how much physical activity the participants usually have, and other characteristics during pregnancy. When their babies are born, the investigators will evaluate the brain development of their babies use magnetic resonance imaging (during natural sleep) at age two weeks and again at age 1&2 years. The investigators will also measure the neurodevelopmental outcomes at age 2 years. Then compare the findings to see if there are group differences in these measures between babies born to normal-weight and obese mothers, if other parameters measured at pregnancy also play a role, and if inflammation markers during pregnancy strongly correlate with infant brain development and neurodevelopmental outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* 11-13 weeks of gestation -≥18 years of age.

Exclusion Criteria:

* BMI measured at first study visit <18.5 or between 26-29 or >50
* hypertension, diabetes, or other preexisting medical conditions known or suspect (by the research team) to influence fetal growth;
* family history of psychological or neurogenetic disorders as determined by the research team that may increase the risk of adverse neurodevelopmental outcomes in offspring
* medications known to influence fetal growth
* recreational drugs, nicotine or tobacco (including smokeless) use or alcohol use while pregnant
* medical conditions developed during pregnancy (e.g. gestational diabetes, preeclampsia) known or suspected by the research team to influence fetal growth
* infants born preterm (<37 weeks of gestation), with congenital defects, intrauterine growth restriction, small for gestational age, macrosomia, hypoglycemia, low Apgar score (<7), or any other medical complications at birth suspected affecting development

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will recruit 260 pregnant women (N=130 for normal weight, BMI 18.5-25, and N=130 for obese, BMI 30-50) at <12 weeks of pregnancy. This is an increase of sample size from the previous number of 120 normal weight women and 120 obese women. The reason is that due to a pandemic, a series factors (such as suspension of all clinical research visits; participants skipping research visits because of COVID concerns) have resulted in that we were not able to get complete data from some of the enrolled subjects at some time points. Our goal is still to obtain complete neuroimaging and maternal clinical data from 120children (N=60/60 from normal-weight or obese mothers) at age ~2 years. .
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2019-10-03 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
To detect changes in brain development by magnetic resonance imaging (MRI) | MRIs will be performed on babies at 2 weeks, 1 year, and 2 years.
  The primary aim is to compare brain development in babies born to lean and obese.mothers by performing MRI scans on babies at 2 weeks, 1 year, and 2 years of life. Mother's BMI will be determined during the clinical visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-10-17): https://cdn.clinicaltrials.gov/large-docs/40/NCT04274140/Prot_ICF_000.pdf